CLINICAL TRIAL: NCT00713492
Title: Computer-Assisted Self-Administration of Ethanol (CASE) in Humans
Brief Title: Computer-Assisted Self-Administration of Ethanol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 080178; 08-AA-0178
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-10-23

CONDITIONS: Alcoholic Intoxication
Keywords: Alcohol; SELF-ADMINISTRATION; Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Alcohol
  Interventions: Drug: Alcohol

INTERVENTIONS:
Drug: Alcohol — human laboratory alcohol consumption.

SUMMARY:
This study will test the reliability of a procedure for self-administering ethanol (alcohol) intravenously (through a vein), using a computer-assisted method. People ordinarily self-administer alcohol through drinking alcoholic beverages, but blood alcohol levels resulting from drinking vary greatly among individuals. For research on alcohol dependence and treatment, a tool for achieving precise blood levels is needed. In addition to testing this method of alcohol administration, the study will examine self-administration behavior and resulting breath alcohol concentration, the effects of alcohol on the participants, and differences between men and women in alcohol self-administration.

Healthy normal volunteers between 21 and 45 years of age may be eligible for this study. Participants are assigned to one of two study groups. Group 1 undergoes three 7-hour study sessions and group 2 participates in two sessions, each of which includes the following procedures:

* Breathalyzer and urine tests for alcohol and illicit drug use.
* Urine pregnancy test for women.
* Light lunch.
* Questionnaire about health and recent drinking.

Alcohol infusion: Subjects are seated in a comfortable chair and instructed on how to use a computer to give themselves a short infusion of alcohol through a catheter (plastic tube) that has been inserted into a vein in their the arm. Sensors are placed on their chest to monitor heart beat and their neck to record skin blood flow. At the start of the session, subjects complete questionnaires about any drug effects and urges to drink they may be feeling. They are trained on how to use the computer to administer alcohol and are then allowed to self-administer alcohol through the catheter any time they like, as long as their peak breath alcohol level does not exceed 0.1 g% (a level that would result from ingestion of 4 to 6 drinks in most people). If that point is reached, the computer automatically inactivates self-administration until the level is lowered again. Breathalyzer readings are taken every 15 to 30 minutes. Subjects may read, watch television or videos or listen to music during the sessions.

Recovery: At the end of the 2.5 hours of self-administration, the catheter is removed and subjects can eat, read, watch television and relax in the clinic until their breath alcohol level falls below 0.02 g%, usually after 2.5 to 3 hours, when they can go home by taxi or with a pre-arranged designated driver.

DETAILED DESCRIPTION:
Objective: The goal of this project is to characterize the computer-assisted self-administration of ethanol (CASE) paradigm by assessing intravenous (IV) alcohol self-administration behavior and the resulting breath alcohol concentration (BrAC) exposure and pharmacologic responses in humans. The study will also evaluate the test-retest reliability of alcohol self-administration and examine the influence of sex and recent drinking history, as well as the effect of acute stress cues on alcohol self-administration. Additionally, this study will test whether a novel experimental paradigm can be used to evaluate impaired control in

heavy drinkers.

Study population: Participants will be 21-60 year-old male and female social drinkers, binge drinkers and heavy drinkers in good health, as determined by medical history, physical exam, ECG and lab tests. Participants with Axis-I psychiatric illness (other than alcohol use disorder for Group 6) will be excluded.

Design: The CASE system utilizes a model-based algorithm based on previously published methods to achieve and maintain pre-determined BrACs using IV alcohol infusions. The CASE system provides flexibility to participants in choosing when to push a button to receive alcohol, as well as flexibility to investigators in controlling the subsequent BrAC exposure. The CASE system allows the investigator to specify and assure the same BrAC increment across all participants, and is set up to prevent the BrAC from exceeding any pre-set upper limit (e.g., 120 mg%).

Following screening, participants will undergo IV ethanol self-administration sessions. Participants will be enrolled in six groups: Group 1 will consist of the first 10 participants who will participate in 3 self-administration sessions (a training session followed by 2 test sessions) to assess the test-retest reliability of alcohol self-administration behavior. Group 2 will consist of 50 participants, who will each participate in 2 self-administration sessions (a training session followed by a test session). During each session, participants will first undergo a directed priming period, lasting 25 min, where they will be prompted to push a button to receive small standardized alcohol infusions. This will be followed by an ad-lib period, lasting up to 2 hrs, where they will have free access to standardized IV alcohol infusions. During the session, BrAC will be measured, heart-rate will be continuously recorded, and subjective perceptions of alcohol effects and urges will be assessed. Group 3 will consist of 15 participants, who will undergo two identical progressive work self-administration sessions for evaluation of test-retest reliability. During each progressive ratio (PR) schedule session, participants will be required to push the button progressively higher number of times for each subsequent alcohol infusion over a 2.5 hr period. Group 4 will consist of 100 participants, who will each participate in 2 sessions: one ad lib self-administration session and one PR schedule self-administration session. Group 5 will consist of 40 participants, who will undergo a baseline self-administration session followed by an interview session for construction of guided imagery scripts. Following this, participants will undergo three alcohol self-administration sessions, following exposure to personalized stress-, alcohol- or neutral-condition associated scripts, presented in randomized order on separate days. Group 6a will consist of a maximum of 15 participants who will undergo a baseline self-administration session followed by an experimental session in which they will be given the opportunity to resist receiving self-infusions of alcohol in return for monetary reinforcers. Group 6b will consist of 37 participants who will complete a baseline self-administration session followed by two experimental sessions, with and without a priming dose of alcohol, and two follow up visits. Group 6 participants will also be given an ecological momentary assessment (EMA) device and will complete random assessments of real-world measures of impaired control and alcohol consumption per day for the duration of the study.

Outcome measures: The primary endpoint is the BrAC exposure (highest BrAC, average BrAC, area-under-the-BrAC-time-curve) achieved during the self-administration session. Additionally, changes in subjective perceptions of alcohol effects, as well as changes in heart rate will be evaluated. The influence of sex and recent drinking history as well as genetic polymorphisms on the self-administration of alcohol will also be examined. Furthermore, individual-specific cellular responses to alcohol exposure will be examined using induced pluripotent stem cells (iPSCs) from participants selected based on genotypic and phenotypic variation in self-administration measures. Outcome measures for group 5 will include stress and alcohol cue-induced craving and self-administration. Human laboratory outcome

measures for Group 6 will include time to lapse during the delay phase, number of infusions,

peak BrAC, and average BrAC during the ad-libitum phase. EMA outcomes will include

total alcohol consumption, number of impaired control episodes, and severity of impaired

control episodes. The CASE paradigm can be a valuable tool for evaluating determinants that may underlie self-administration behavior in humans. The effect of pharmacological agents on alcohol self-administration can be evaluated as a marker of the clinical effectiveness of these agents in the treatment of alcohol-dependence.

ELIGIBILITY:
* GROUPS 1-5:

All participants will be between the ages of 21 and 45 years, social drinkers in good health. Young females will have normal menstrual cycles and will be tested during the follicular phase of their cycle (within 10 days of offset of menses) and must have a negative urine pregnancy (hCG) test at the start of the study session.

INCLUSION CRITERIA:

1. Male and female participants between 21-45 years of age.
2. Good health as determined by normal or non-clinically-significant findings on medical history, physical exam, ECG and lab tests.
3. Female participants will be tested during the follicular phase of their cycle (within 10 days of offset of menses) and must have a negative urine pregnancy (hCG) test at the start of each study session. For Group 5, due to the number of study visits, female subjects will be tested outside the menses phase of their cycle.
4. Group 5 will include 20 subjects who report at least 2 binge drinking episodes in the month prior to the study (a binge episode is defined as consuming at least 4 drinks for females and at least 5 drinks for males during the drinking episode) and 20 subjects

who report no binge drinking episodes in the past month.

EXCLUSION CRITERIA:

1. Current or prior history of serious medical illness, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders.
2. Positive hepatitis A, B antigen or C or HIV test at screening.
3. Current history of Axis-I psychiatric illness.
4. Current or lifetime diagnosis of alcohol or substance dependence.
5. Currently seeking treatment for alcohol use disorders.
6. History of significant withdrawal symptoms or presence of clinically significant withdrawal symptoms (Clinical Institute Withdrawal Assessment (CIWA) score > 8) at screening.
7. Non-drinkers (alcohol-na(SqrRoot) ve individuals or current abstainers) or individuals with no experience drinking 5 or more drinks on one occasion in their lifetime.
8. Regular tobacco users will be excluded from the study in order to avoid nicotine withdrawal symptoms. Occasional use of tobacco products (up to 20 cigarettes/week) is acceptable. For Groups 3, 4 and 5, participants must be current non-smokers (past smokers who have quit for over 1 year can be included).
9. Positive result on urine drug screen or positive breathalyzer during screening visit or at the start of any study visit.
10. Pregnancy or intention to become pregnant for women. Female participants will undergo a urine beta-hCG test to ensure they are not pregnant.
11. Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and

    ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, and narcotics including propoxyphene, oxycodone and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Cough-and-cold preparations which contain anti-histamines, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, should be withheld for at least 72 hours prior to each study session.
12. Current or prior history of alcohol-induced flushing reactions.
13. Female participants who have abnormal menstrual cycles in the absence of irregularities caused by hormonal contraception, as defined by irregularities in menstrual cycle length (cycles of >36 days or < 8 cycles per year), clinically significant menstrual periods that are heavier or lighter than usual, and/or accompanied by significant pain, cramping or nausea and vomiting that requires intervention.

GROUP 6

Group 6 will include heavy drinkers between the ages of 21 and 60 years, in good health. Unfortunately, heavy drinking does not have a universally agreed upon definition and the criteria used to define heavy drinking vary from study to study. There is evidence that

incorporating both amount of alcohol consumed per occasion and amount of alcohol consumed per week is relevant to account for risk related to pattern of drinking and total consumption. Therefore in our study we will select heavy drinkers using a definition that takes into account both pattern of drinking and total consumption. For pattern of drinking, we will require our subjects to have on average at least one binge drinking day per week, using the NIAAA definition of 5 or more drinks for men and 4 or more drinks for women (NIAAA website). For total consumption, we will use an average of 8 or more drinks per week for women and 15 or more drinks per week for men as this level of drinking has been shown to confer increased risk of mortality.

INCLUSION CRITERIA:

1. Male and female participants between 21-60 years of age.
2. Male participants must have consumed an average of 15 or more standard drinks per week and females must have consumed an average of 8 or more standard drinks per week during the past 90 days. Average number of drinks per week will be calculated based on total number of drinks as measured by the timeline followback (TLFB) (e.g., for 90 days worth of data, total drinks divided by 90 and then multiplied by 7 will be the average number of drinks per week).
3. Participants must have on average at least 1 binge drinking day per week during the last 90 days, defined as a day in which 4 or more standard drinks were consumed for females and 5 or more standard drinks were consumed for males. Average number of binge drinking days will be calculated based on total number of binge drinking days from the TLFB (e.g. for 90 days worth of data, participants with a total of 13 or more binge drinking days will be eligible).
4. Participants must be able and willing to refrain from consuming alcohol 24 hours prior to each alcohol self-administration session.

EXCLUSION CRITERIA:

1. Current or prior history of serious medical illness, including CNS, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders.
2. Positive hepatitis A, B antigen, or C or HIV test at screening.
3. Abnormal findings on ECG, unless cleared for participation by cardiologist or Licensed Independent Practitioner (LIP).
4. Current history of major depressive disorder, bipolar disorder, psychotic disorder, obsessive compulsive disorder (OCD), post-traumatic stress disorder (PTSD), eating disorder, or any other Axis-I psychiatric disorders requiring intervention.
5. An aspartate transaminase (AST) or alanine transaminase (ALT) level more than 3 times the upper limit of normal.
6. Current (past 12 months) diagnosis of substance use disorder other than alcohol use disorder, unless in early remission (no criteria met for at least 3 months).
7. Positive result on urine drug screen or breathalyzer test during initial or update visit under the screening protocol (14-AA-0181) most proximal to enrollment. Positive urine drug screen during more than 1 study visit or breathalyzer reading during more than 1 self-administration study visit will result in participant withdrawal from the study.
8. Currently seeking treatment for alcohol use disorder or having undergone inpatient or outpatient detoxification or treatment for alcohol problems in the past 6 months.
9. History of significant withdrawal symptoms or presence of clinically significant withdrawal symptoms (Clinical Institute Withdrawal Assessment (CIWA) score > 8) at screening.
10. Pregnancy, intention to become pregnant, or breastfeeding. Female participants will undergo a urine beta-hCG test to ensure that they are not pregnant.
11. Medication exclusion criteria:

    1. . Daily or regular use of prescription or OTC medications known to interact with alcohol in the 2-week period prior to assessment. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, anti-epileptics including phenytoin and phenobarbital codeine, and narcotics including propoxyphene, oxycodone and hydrocodone.
    2. Daily or regular use of drugs known to inhibit or induce enzymes that metabolize alcohol in the 4-week period prior to assessment. These include chlorzoxazone, isoniazid, metronidazole and disulfiram. Note that any discontinuation of medications will only be done at the recommendation of a physician.
12. Current or prior history of alcohol-induced flushing reactions.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2008-10-29 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
BrAC Exposure (peak BrAC, Average BrAC) during self-administration | 2.5 hrs
  alcohol consumption measured during human lab session.

SECONDARY OUTCOMES:
Subjective response during self-administration | 2.5 hrs
  alcohol consumption measured during human lab session.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Sloan ME, Grant CW, Stangl BL, Klepp TD, Brewton HW, Cinar R, Kunos G, Ramchandani VA. The effects of acute alcohol administration on circulating endocannabinoid levels in humans. Addict Biol. 2022 Sep;27(5):e13197. doi: 10.1111/adb.13197. PMID 36001429
- [Derived] Vatsalya V, Stangl BL, Ramchandani VA. Assessment of Skin Blood Flow Following Acute Intravenous Alcohol, and Association with Subjective Perceptions, in Social Drinkers. Alcohol Clin Exp Res. 2019 Mar;43(3):405-410. doi: 10.1111/acer.13962. Epub 2019 Feb 8. PMID 30735255
- [Derived] Gowin JL, Sloan ME, Stangl BL, Vatsalya V, Ramchandani VA. Vulnerability for Alcohol Use Disorder and Rate of Alcohol Consumption. Am J Psychiatry. 2017 Nov 1;174(11):1094-1101. doi: 10.1176/appi.ajp.2017.16101180. Epub 2017 Aug 4. PMID 28774194
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-AA-0178.html